CLINICAL TRIAL: NCT05916196
Title: [18F]FLUOROESTRADIOL (FES) PET/CT IMAGING OF THE ESTROGEN RECEPTOR IN PATIENTS WITH METASTATIC OR RECURRENT UTERINE CANCER
Brief Title: [18F]FES PET/.CT in Uterine Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 852782; UPCC 30822 (Other: ACC)
Record Dates: First submitted 2023-04-18; First posted 2023-06-23 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Uterine Cancer
Keywords: estrogen receptor PET imaging
MeSH Terms: conditions — Uterine Neoplasms | interventions — 16-fluoroestradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Recurrent or metastatic uterine cancer (Experimental): Women with known or suspected recurrent or metastatic uterine cancer may be eligible for this study. Patients may participate in this study if they are at least 18 years of age, most participants will be receiving care at the clinical practices of the University of Pennsylvania.
  [18F]fluoroestradiol (FES) PET/CT imaging will be used to evaluate estrogen receptor (ER) activity in areas of disease known by standard of care imaging (e.g. CT, MRI, Bone Scan, FDG PET/CT, ultrasound) or clinical exam. For patients starting a new line of therapy, imaging will occur prior to starting new therapy. For patients who completed an initial scan and are starting new therapy, some patients may also undergo a second FES PET/CT scan at the time of suspected progression of disease to compare for changes in FES uptake measures (prior to initiation of next line therapy).
  Interventions: Drug: 18F-Fluoroestradiol

INTERVENTIONS:
Drug: 18F-Fluoroestradiol — 18F-FES PET/CT
  Other Names: 18F-FES

SUMMARY:
Women with known or suspected recurrent or metastatic uterine cancer may be eligible for this study. Patients may participate in this study if they are at least 18 years of age, most participants will be receiving care at the clinical practices of the University of Pennsylvania.

[18F]fluoroestradiol (FES) PET/CT imaging will be used to evaluate estrogen receptor (ER) activity in areas of disease known by standard of care imaging (e.g. CT, MRI, Bone Scan, FDG PET/CT, ultrasound) or clinical exam. For patients starting a new line of therapy, imaging will occur prior to starting new therapy. For patients who completed an initial scan and are starting new therapy, some patients may also undergo a second FES PET/CT scan at the time of suspected progression of disease to compare for changes in FES uptake measures (prior to initiation of next line therapy). The selection of therapy will be made by a treating physician and will not be affected by participation in this imaging study. Results of the FES PET/CT scan may be shared with the treating physician or subject by request but will not be used to make clinical decisions about treatment.

DETAILED DESCRIPTION:
This is a phase II study using the novel radiotracer [18F]fluoroestradiol (FES). Patients with metastatic, recurrent, or intact non-operated uterine cancer not treated with surgery. Patients may participate in this study if they are at least 18 years of age. Volunteers that meet the eligibility criteria will be considered for study participation regardless of race or ethnic background. We anticipate enrolling up to 30 evaluable subjects who meet eligibility requirements for this study, due to the nature of the disease population all subjects will be women. Subjects will be considered evaluable if they complete at least one FES PET/CT scan. Patients who come to the University of Pennsylvania for diagnosis and/or treatment of this gynecological cancer may be approached by study personnel for recruitment into this study. Patients will be approached initially in person, by phone or email about study participation. After discussion of the study procedures, risks and benefits, if the subject agrees to participate in the study, the FES PET/CT will be ordered by a physician and scheduled. Subjects may cancel the scan appointment at any time prior to the injection of FES with no negative impact to them or their medical care at University of Pennsylvania. A written informed consent will be reviewed with the subject and signed prior to any study procedures being performed. The selection of therapy will be made by a treating physician and will not be affected by participation in this imaging study.

Accrual will likely occur over approximately 2 years. Subjects who are enrolled but are unable to complete the entirety of their FES imaging procedure will be considered non-evaluable. If this occurs, we will plan to replace this subject in the enrollment, due to this we anticipate that we may enroll up to 40 subjects in order to meet our target enrollment of 30 evaluable subjects.

Participants will undergo up to two FES PET/CT scans. The first scan is the initial study scan and the only required of the study. A second optional FES PET/CT scan may be done at the time of progression after initiation of therapy, prior to initiation of next line therapy, to collect data on the changes in FES uptake with therapy and therapy utilized.

Positron emission tomography (PET) imaging will be used to evaluate estrogen receptor activity in sites of metastatic uterine cancer using the investigational radiotracer [18F]FES. Imaging will be performed using a whole-body PET/CT scanner. The protocol will be performed under the regulatory approval of the IRB and FDA IND. Subjects will undergo a skull base to mid-thigh PET/CT scan starting at approximately 60 minutes after [18F]FES injection. Images will be reconstructed using standard reconstruction techniques.

If a patient will be undergoing a clinical biopsy or surgery, they may be asked to consent for collection of tissue for the purposes of this research study. If the investigator deems that there is a site accessible for research biopsy, the subject may be consented for an optional research only biopsy at baseline and after starting treatment; however, consent for research tissue collection is not required for entry into the study. Results of standard uterine cancer pathology immunohistochemistry (IHC) which includes estrogen receptor (ER), will be collected from archival tissue if available and performed on any new biopsy.

A research blood sample may be collected at the time of the FES PET/CT scan that will be evaluated for the presence of circulating tumor cells (CTCs) and circulating tumor DNA (ctDNA). Identified CTCs will be tested for estrogen receptor positivity. Serum estradiol and other related levels including sex hormone-binding globulin (SHBG) will be analyzed. FES uptake measures will be compared to the number of ER+ CTCs and the ratio of ER + to ER- CTCs present. This blood draw will be optional and may be omitted at the choice of the investigator or the subject

ELIGIBILITY:
Inclusion Criteria

1. Participants will be ≥ 18 years of age
2. Recurrent or metastatic or intact non-operated uterine cancer not treated with surgery that is biopsy-proven or demonstrated on other standard of care imaging (e.g. CT, FDG PET/CT, MRI, bone scan, x-ray, ultrasound)
3. At least one lesion outside the liver detected by standard of care imaging (e.g.CT, FDG PET/CT, MRI, bone scan, x-ray, ultrasound)
4. Participants must be informed of the investigational nature of this study and be willing to provide written informed consent and participate in this study in accordance with institutional and federal guidelines prior to study-specific procedures.
5. Subjects that are currently on or have recently discontinued tamoxifen or fulvestrant would require an 8-week or 28-week, respectively, washout period prior to FES PET/CT scan.

Exclusion Criteria

1. Females who report they are pregnant at screening will not be eligible for this study. A urine pregnancy test will be performed in women of child-bearing potential prior to FES injection.
2. Inability to tolerate imaging procedures in the opinion of an investigator or treating physician
3. Any current medical condition, illness, or disorder as assessed by medical record review and/or self-reported that is considered by a physician investigator to be a condition that could compromise participant safety or successful participation in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Uterine cancer is only possible in women who were born female
Enrollment: 30 (Estimated)
Dates: Start 2024-04-05 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
rate of FES positivity in ER+ uterine cancer | 1 year
  Evaluate utility of FES PET/CT to detect estrogen receptor (ER+) uterine cancer lesions in patients with recurrent or metastatic uterine cancer

SECONDARY OUTCOMES:
Number of FES positive sites compared to standard of care imaging | 6 weeks
  Evaluate utility of FES PET/CT compared to standard axial cross-sectional imaging and/or FDG PET/CT when available to establish tumor heterogeneity and staging
PFS | 5 years
  Correlate FES uptake with estimate of progression-free survival
Pathology | 6 weeks
  Correlate FES PET/CT uptake measures with standard and experimental pathology (e.g. estrogen receptor-alpha, estrogen receptor-beta)
Change in FES at progression | 1 year
  In patients who receive a second FES PET/CT scan, compare FES uptake in patients at initial scan and at progression

CONTACTS AND LOCATIONS:
Overall Officials: Neil Taunk, MD, Principal Investigator — Abramson CC
Locations (1):
- Abramson Cancer Center at University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No